CLINICAL TRIAL: NCT01789619
Title: Extended Release Tacrolimus (Advagraf®) in Severe Adult Atopic Dermatitis Patients
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr M.S. de Bruin-Weller, MD, PhD, UMC Utrecht
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extended release tacrolimus (Advagraf®)
  Interventions: Drug: Extended release tacrolimus (Advagraf®)

INTERVENTIONS:
Drug: Extended release tacrolimus (Advagraf®)

SUMMARY:
To evaluate the clinical efficacy of the extended release formulation of tacrolimus (Advagraf®) in patients with severe atopic dermatitis, who can not be treated adequately with cyclosporine A because of side effects and/or non-responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe atopic dermatitis, uncontrolled by topical treatment (indication for oral immunosuppressive drugs), who are unresponsive to Cyclosporin A, or in which treatment was discontinued because of side effects.

Exclusion Criteria:

* Concomitant use of other oral immunosuppressive drugs and/or UV light therapy
* Preexisting abnormalities in liver function, kidney function or haematological abnormalities
* History of malignancy within the last 5 years
* Uncontrolled hypertension
* Pregnancy or lactation; wish for pregnancy during the treatment period
* Infections requiring continued therapy
* Known positivity for HIV
* Evidence of drug and/or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe atopic dermatitis, who can not be treated adequately with Cycloporin A because of side effects and/or non-responsiveness.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Scoring Atopic Dermatitis (SCORAD) | Every 4 weeks up to one year
  Clinical eczema scores

SECONDARY OUTCOMES:
Change in Patient-Oriented Eczema Measure (POEM) | Every 4 weeks up to one year
  Self administered eczema score
Change in Thymus and Activation-Regulated Chemokine in serum (TARC) | Every 4 weeks up to one year
  Biomarker atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: C AFM Bruijnzeel-Koomen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands